CLINICAL TRIAL: NCT02032147
Title: Treatment of Cerebral Radiation Necrosis (CRN) With Nerve Growth Factor (NGF)
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fan Ming, MD,PhD, Fudan University
Other Study IDs: CRN2009
Record Dates: First submitted 2013-09-27; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Cerebral Necrosis; Nashopharyngeal Cancer; Nerve Growth Factor
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- NGF group: This group will be treated with NGF 18u daily for 60 days.
  Interventions: Drug: NGF group
- control group: this group will receive conservative therapy such as hyperbaric therapy or corticosteroids therapy or "wait and see" policy

INTERVENTIONS:
Drug: NGF group — This group will be treated with NGF 18u per day im for 60 days
  Groups: NGF group

SUMMARY:
Cerebral radiation necrosis (CRN) is a well-documented late complication of radiation therapy for cancers, and may have a devastating effect on the patient's quality of life (QOL). However,CRN was once regarded as a progressive and irreversible disease, no standard therapy has been suggested for CRN. In our clinical practice, we have used nerve growth factor(NGF) to treat CRN, and found that GM1 can successfully reverse CRN. A case report has been published in Journal of Clinical Oncology (JCO) in 2011. So we carried out this prospective study to test the efficacy of NGF for CRN.

ELIGIBILITY:
Inclusion Criteria:

* The necrotic mass shown on MRI must be measured in two dimensions. No local or regional recurrence, no distant metastasis. Karnofsky performance status of at least 70 and were supposed to live more than 6 months.

Exclusion Criteria:

* CRN combined with local or regional relapse, or with distant metastasis.
* CRN combined with other cerebrovascular disease.
* CRN combined with the second primary malignancy.
* CRN without neurologic symptoms or signs.
* CRN combined with diabetes.
* CRN patients that were supposed to live less than 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have undergone definitive RT for histologically confirmed NPC years before. They were required to have at least two consecutive magnetic resonance imaging (MRI) study supporting the diagnosis of CRN with an interval of 3-4 months, with the second MRI showing progressive disease compared with the first MRI. The necrotic mass shown on MRI must be measured in two dimensions in order to define the response to treatment. Other radiologic studies were also required to support the non-existence of local or regional recurrence, distant metastasis. Patients must have undergone mental status examinations and had progressive neurologic symptoms or signs. In addition, they were required to have a Karnofsky performance status of at least 70 and were supposed to live more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
efficacy of using NGF for treating CRN | 6-8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China